CLINICAL TRIAL: NCT04188899
Title: Point-of-care Ultrasound in the Assessment of Snake Bite
Status: Recruiting | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: 1910093637
Record Dates: First submitted 2019-12-02; First posted 2019-12-06 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Rattlesnake Bite (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early identification of tissue injury from a rattlesnake bite is critical to prevent complications and reduce health care costs. Given the limitations of clinical assessment, there is a need to develop a more objective reproducible, anatomically detailed diagnostic tool for to accurately assess tissue damage and assist with timely administration of antivenom, if needed. Emergency physician performed point-of-care ultrasonography has been shown to be beneficial in the diagnosis and management of skin and soft tissue infections. The innovative use of bedside ultrasound technology can provide new information to individualize antivenom treatment and to improve patient outcomes. The objectives of this study is to compare clinical assessment and bedside ultrasound findings in the detection of tissue injury in emergency department patients with rattle snakebite and determine if bedside ultrasound can alter management (antivenom dosing) in emergency department patients with rattle snakebite.

DETAILED DESCRIPTION:
Arizona has the highest per capita rate of rattlesnake envenomation (the process by which venom is injected by the bite of a venomous animal) in the United States leading to millions of dollars in health care costs. Local tissue destruction typically manifests in the first few hours after snakebite and can progress over days or weeks leading to long-term complications such as muscle, nerve, and circulatory damage. The cornerstone in the treatment of rattlesnake envenomation is accurate estimation of progression of local tissue damage and timely administration of antivenom to halt the progression of venom effects. The initial decision to administer antivenom is based on clinical parameters such as edema, induration, bullae and blisters. The need for repeat doses of antivenom is determined by serial clinical assessments and laboratory parameters. However, no definitive clinical or laboratory parameters currently exist. The current practice is limited by inter-observer variability in the clinical assessment and the inability to accurately assess the extent of tissue injury. In a significant number of cases, it is difficult to accurately track the progression of the venom effects until they become more pronounced and severe. With the limitations of clinical assessment, administration of antivenom is delayed potentially resulting in poor patient outcomes. A further complicating factor is that not all rattlesnake bites result in envenomation. A substantial number of bites by rattlesnakes can result in "dry bite" in which snake venom is not transferred from snake to human and thus will not cause tissue destruction.4 Because of limitations of clinical assessments, these patients receive antivenom even though it is not necessary. This liberal and inappropriate use of antivenom is not cost effective and can also affect patient safety.

Early identification of tissue injury from a rattlesnake bite is critical to prevent complications and reduce health care costs. Given the limitations of clinical assessment, there is a need to develop a more objective reproducible, anatomically detailed diagnostic tool for to accurately assess tissue damage and assist with timely administration of antivenom, if needed. Emergency physician performed point-of-care ultrasonography has been shown to be beneficial in the diagnosis and management of skin and soft tissue infections. The innovative use of bedside ultrasound technology can provide new information to individualize antivenom treatment and to improve patient outcomes. The quick, noninvasive nature and repeatability of point-of-care ultrasonography makes it an ideal objective tool for the assessment of emergency department (ED) patients with rattle snakebites. Ultrasound technology can reveal subcutaneous edema, localized fluid collections, tissue necrosis, and muscle contractions resulting from a rattlesnake bite.6 Point-of-care ultrasonography performed by emergency physicians can detect the tissue injury that is not evident on clinical assessment and accurately track the patterns of injury prior to their external manifestations. This innovative approach can expedite treatment in patients with rattle snake envenomation thereby preventing complications such as coagulopathy (a condition in which the blood's ability to clot is impaired) and compartment syndrome (excessive pressure build up inside an enclosed space in the body). Additionally ultrasound can eliminate the inappropriate use of antivenom in patients with dry bite potentially reducing health care costs and improving patient safety.

Our preliminary experience and prior literature suggests that point-of-care ultrasound can detect subcutaneous edema, help clinicians to make an accurate assessment of proximal progression of local findings due to a snake bite and can expedite the consultation and appropriate treatment in patients with snake bite.The objectives of this study is to compare clinical assessment and bedside ultrasound findings in the detection of tissue injury in emergency department patients with rattle snakebite and determine if bedside ultrasound can alter management (antivenom dosing) in emergency department patients with rattle snakebite.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older)
* Both genders
* Complaint of snake bite

Exclusion Criteria:

* If they are unwilling to provide informed consent
* Hemodynamically unstable patients (shock respiratory distress, altered mental status, and cardiorespiratory arrest)
* All vulnerable patient populations, e.g., children, pregnant patients, prisoners, and patients unable to verbally consent due to cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patients presenting with Rattle snake envenomation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants in whom ultrasound detected progress of skin changes earlier than physical examination | First 10 hours of Emergency Department encounter
  Sonographic skin changes

CONTACTS AND LOCATIONS:
Overall Officials: Srikar Adhikari, MD, MS, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center-Tucson, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided